CLINICAL TRIAL: NCT06787833
Title: The Effect of Performing Clinical Practice with Classical Music on Dental Students' Stress and Anxiety During the COVID-19 Pandemic
Brief Title: The Effect of Classical Music on Dental Students' Stress and Anxiety During the COVID-19 Pandemic
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karabuk University (Other)
Collaborators: Ankara University (Other)
Responsible Party: Principal Investigator, Sevilay Yeğinoğlu, Department of Periodontology, Principal Investigator, Asst. Prof. Dr., Karabuk University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: No.17/03, dated 17.11.2021
Record Dates: First submitted 2025-01-16; First posted 2025-01-22 (Actual); Last update posted 2025-01-22 (Actual); Status verified 2025-01

CONDITIONS: Psychological Factors
Keywords: Beethoven; Coronavirus anxiety; Music; Mozart; Perceived stress
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Participants (Experimental): they were asked to complete a questionnaire including socio-demographic data, Perceived Stress Scale (PSS-14), and Coronavirus Anxiety Scale (CAS) before patient admission (T1). The students were asked to complete the same questionnaire at the end of the day after working for 2 days (T2) and in the morning on the 5th day of their study before seeing patients (T3). Each of the students participating in the study was given disposable headphones every day during the week of music listening. In this study, Beethoven's Moonlight Sonata (1 hour 2 minutes), Mozart's Serenata Notturna KV239 (12.50 minutes) and Pachelbel's Canon in D major (6.16 minutes) were used. It was shared with the students via WhatsApp and they were allowed to listen to this music on their phones for 1 week (2 hours on average) during the study period. The same questionnaire was refilled at the end of the week in which music was played (T4).
  Interventions: Other: Questionnaire; Other: listening to music

INTERVENTIONS:
Other: Questionnaire — to complete a questionnaire including socio-demographic data, Perceived Stress Scale (PSS-14), and Coronavirus Anxiety Scale (CAS) before patient admission (T1). The students were asked to complete the same questionnaire at the end of the day after working for 2 days (T2) and in the morning on the 5th day of their study before seeing patients (T3).The same questionnaire was refilled at the end of the week in which music was played (T4).
Other: listening to music — Each of the students participating in the study was given disposable headphones every day during the week of music listening. In this study, Beethoven's Moonlight Sonata (1 hour 2 minutes)23,55, Mozart's Serenata Notturna KV239 (12.50 minutes)18,19, and Pachelbel's Canon in D major (6.16 minutes)24,25 were used. It was shared with the students via WhatsApp and they were allowed to listen to this music on their phones for 1 week (2 hours on average) during the study period.

SUMMARY:
The students adapted to the environment for the first 2 days, were informed about the study, and their informed consent was obtained. Participants were asked to answer all questions and to give a single answer to each question. The students filled in the questionnaire form used in the study without any intervention by the researcher. Participants filled out the same survey four times at different times following a specific protocol.

DETAILED DESCRIPTION:
The study was conducted with a specific protocol. First, they were asked to complete a questionnaire including socio-demographic data, Perceived Stress Scale (PSS-14), and Coronavirus Anxiety Scale (CAS) before patient admission (T1). The students were asked to complete the same questionnaire at the end of the day after working for 2 days (T2) and in the morning on the 5th day of their study before seeing patients (T3). Each of the students participating in the study was given disposable headphones every day during the week of music listening. In this study, Beethoven's Moonlight Sonata (1 hour 2 minutes) Mozart's Serenata Notturna KV239 (12.50 minutes) and Pachelbel's Canon in D major (6.16 minutes)were used. It was shared with the students via WhatsApp and they were allowed to listen to this music on their phones for 1 week (2 hours on average) during the study period. The same questionnaire was refilled at the end of the week in which music was played (T4).

ELIGIBILITY:
Inclusion Criteria:

* Aged 20 years and over,
* Systemically healthy and drug-free,
* Students who were obliged to practice in the clinic of the Department of Periodontology, Faculty of Dentistry, Ankara University, within the scope of the education program

Exclusion Criteria:

* Systemic diseases
* Medication use

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2021-11-01 (Actual); Primary Completion 2021-12-17 (Actual); Study Completion 2021-12-24 (Actual)

PRIMARY OUTCOMES:
Participants' initial stress and anxiety levels | up to 2 days
  In the period after the transition from remote learning to face-to-face education during the pandemic, it was determined that final-year dental students engaged in clinical practice experienced moderate levels of perceived stress and low levels of coronavirus anxiety.

SECONDARY OUTCOMES:
Participants' stress and anxiety levels after listening to music | up to 2 weeks
  In this situation, the music played to the students was effective, as declines were observed in survey scores. However, relaxation and breathing exercises could also be recommended to dental students, who experience a stressful education process even outside of the pandemic. Psychological support and counseling could be provided when necessary.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Karabuk University, Karabük, Karabük Province
  - AnkaraUniversity, Ankara

IPD SHARING:
Plan to Share IPD: Yes
We can share statistical data in excel file upon request.
Supporting Information: Study Protocol, SAP
Time Frame: Start date: Jan 2025 End date: Jan 2030
Access Criteria: Data sharing can be done when they contact the corresponding author.
URL: https://www.dentistry.ankara.edu.tr/klinik-arastirmalari-etik-kurulu/

REFERENCES:
- [Background] Groarke JM, Hogan MJ. Listening to self-chosen music regulates induced negative affect for both younger and older adults. PLoS One. 2019 Jun 6;14(6):e0218017. doi: 10.1371/journal.pone.0218017. eCollection 2019. PMID 31170224